CLINICAL TRIAL: NCT01356563
Title: Effects of Pharmacist on Medication-related Problems in Hemodialysis Patients: a Randomized,Controlled, Double-blind Study
Brief Title: Efficacy Study of Pharmacist Intervention on Medication-related Problems in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sin-Lau Hospital (Other)
Responsible Party: Chen Hung-Yi, Tainan Sin-Lau Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SLH-100-05
Record Dates: First submitted 2011-05-14; First posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis
Keywords: hemodialysis; pharmacist; medication-related problems; compliance
MeSH Terms: conditions — Patient Compliance | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clinical pharmacist intervention (Experimental)
  Interventions: Behavioral: pharmaceutical care
- usual care (No Intervention): Patients randomized to usual care group will receive routine review of medication by outpatient department pharmacists and nurse.

INTERVENTIONS:
Behavioral: pharmaceutical care — Hemodialysis patients in the intervention group will receive pharmaceutical care delivered by clinical pharmacist, which including personal interview, medication review, medication reconciliation, patient education and recommended actions
  Arms: clinical pharmacist intervention

SUMMARY:
The investigators propose that pharmacist interventions would reduce the amount of unresolved medication-related problems in hemodialysis patients.

Condition:Hemodialysis patients

Intervention:Behavioral,Pharmacist intervention

Study Design:Randomized Allocation

Control: Active Control

Endpoint Classification: Efficacy Study

Intervention Model: Parallel Assignment

Masking: Double Blind (Caregiver, Outcomes Assessor)

Primary Purpose: Treatment

DETAILED DESCRIPTION:
Introduction:

End stage renal disease (ESRD) incidence in Taiwan ranked first and prevalence ranked second in the world from 2002 to 2005. Several foreign researches had reported that hemodialysis (HD) patients often require 12 medications to treat 5 to 6 comorbid conditions. Besides, ESRD is a lifelong disease and rates of compliance may diminish overtime. Thus, HD patients may be at particular risk for drug related problems, durg-drug interactions and noncompliance. Our aim is to analysis the effect of pharmacist in medication-related problems in ambulatory hemodialysis patients.

Methods:

This study is a randomized double-blind, active controlled trial. The investigators will invite and communicate with HD patients to find medication -related problems. After pharmacist evaluation, pharmacist will do pharmaceutical interventions to resolve medication-related problems, drug-drug interactions etc. in experimental group. In the active control group, pharmacist in this study will not do pharmaceutical interventions. The investigators will monitor each patient in a two-week period for medication-related problems.

Our primary outcome is the amount of unresolved medication-related problems in each group after two weeks. Blind outcome assessor will evaluate the amount of unresolved medication-related problems in each case as well as compliance in these patients after two weeks.

The investigators suppose that clinical pharmaceutical intervention will reduce the amount of unresolved medication-related problem in experimental group. On the other hand, patients without clinical pharmaceutical intervention will have more unresolved medication-related problems.

ELIGIBILITY:
Inclusion Criteria:

* 20-96 years old hemodialysis patient taking medications prescribed by nephrologists.

Exclusion Criteria:

* Patients who refused informed consent
* Cognitive impaired
* unable to talk or hearing disability

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-12 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
amount of unsolved medication-related problems in each group | 14 days
  Clinical pharmacist provide pharmaceutical care in experimental group in order to reduce medication-related problems. With pharmaceutical care, we suppose that amount of unsolved medication-related problems will less than the control group.

SECONDARY OUTCOMES:
Patient self-reported medication compliance | 14 days after recruitment
  14 days after recruitment, outcome assessor will record patient self-reported medication compliance. 1 score means almost noncompliance,while 5 score means that patient takes almost every medication.
pharmaceutical care satisfaction | 14 days after recruitment
  From 1 score to 5 scores, 1 score means that patient is very unsatisfied with pharmaceutical care in the past 14 days. 5 scores means that patient is very satisfied with pharmaceutical care in the past 14 days.
adverse events | 14 days after recruitment
  An adverse event is any adverse change in health or side effect that occurs in a person who participates in our clinical trial while the patient is receiving the medications prescribed by physician.
knowledge about medication | 14 days after recruitment
  Patient self-reported knowledge about medication. From 1 score to 5 scores, as the score increase, it means that patients know more information about his medication.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yi Chen, Principal Investigator — Sin-Lau Hospital
Locations (2):
- Taiwan (2):
  - Sin-Lau hospital, Tainan, Tainan
  - Tainan Sin-Lau Hospital, Tainan

REFERENCES:
- [Background] Yang WC, Hwang SJ; Taiwan Society of Nephrology. Incidence, prevalence and mortality trends of dialysis end-stage renal disease in Taiwan from 1990 to 2001: the impact of national health insurance. Nephrol Dial Transplant. 2008 Dec;23(12):3977-82. doi: 10.1093/ndt/gfn406. Epub 2008 Jul 15. PMID 18628366
- [Background] Schmid H, Schiffl H, Lederer SR. Pharmacotherapy of end-stage renal disease. Expert Opin Pharmacother. 2010 Mar;11(4):597-613. doi: 10.1517/14656560903544494. PMID 20163271
- [Background] Manley HJ, Bailie GR, Grabe DW. Comparing medication use in two hemodialysis units against national dialysis databases. Am J Health Syst Pharm. 2000 May 1;57(9):902-6. doi: 10.1093/ajhp/57.9.902. No abstract available. PMID 10840531